CLINICAL TRIAL: NCT04522193
Title: Physiopathology of Dumping Syndrome in Esophageal Atresia
Brief Title: Dumping Syndrome and Esophageal Atresia
Acronym: DUMTORING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other); french patient association for oesophageal atresia AFAO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019_51; 2020-A01938-31 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Oesophageal Atresia; Dumping Syndrome
Keywords: Oesophageal dysmotility; Oesophageal atresia; Post prandial hypoglycaemia; Gastric emptying troubles
MeSH Terms: conditions — Esophageal Atresia; Dumping Syndrome; Esophageal Motility Disorders; Hypoglycemia | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All children born at the Lille University Hospital during the investigation period with esophageal atresia type III or IV
  Interventions: Device: Glycemic Holter; Radiation: gastric emptying scintigraphy; Device: Holter ECG

INTERVENTIONS:
Device: Glycemic Holter — Continuous glycaemia monitoring,
Radiation: gastric emptying scintigraphy — Fasting administration of a Technecium-labelled milk bottle and quantification of the remaining radioactivity by a camera every 30 minutes for 4 hours.
Device: Holter ECG — continuous cardiac monitoring

SUMMARY:
Dumping syndrome (DS) is frequent in oesophageal atresia (29%). In causing hypoglycaemia, it can be dangerous for neonates. Mechanisms of DS are actually partialy understood. This is also an affection difficult to diagnose, because it only occurs after meals and can be inconstantly present. To date, their is only symptomatic treatment for DS. This study aims to understand its pathological mechanisms so as to better treat it and avoid its consequences. Oesophageal atresia patients enrolled in this study will benefit from a continuous glycemic monitoring, a continuous cardiac monitoring, and an a gastric emptying scintigraphy at the age of 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patients operated at birth for Oesophageal atresia type C
* Aged from 2 to 3 months at inclusion
* Off prokinetic treatment (suspended for at least 72 hours) before monitoring

Exclusion Criteria:

* History of dumping syndrome of other cause (microgastria, fundoplication, dysautonomia..)
* History of any disease that can modify glycemic regulation (hyperinsulinism, neonatal diabete)
* Treatment that can modify gastric motility

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Abnormal glycaemia associated with vagal hypertonia | At least once during the 48 hours monitoring
  Composite criteria: association between abnormal glycaemia (high or low) and variations of cardiac frequency

SECONDARY OUTCOMES:
Abnormal glycaemia associated with abnormal gastric emptying | At least once during the 48 hours monitoring
  Composite criteria: association between abnormal glycaemia (high or low) and abnormal gastric emptying study
Persistance of dumping syndrome | At the age of 6 months
  measured by a gastric emptying scintigraphy
Tolerance of glucose monitoring | At least once during the 48 hours monitoring
  Occurrence of side effects or technical issues during monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Madelaine AUMAR, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Hôpital Jeanne de Flandres, Lille
  - Hôpital Jeanne de Flandre - Pôle enfant, CHU de Lille, Lille